CLINICAL TRIAL: NCT00757484
Title: Evaluation of Postoperative Blood Pressure Changes After Benign Gynecologic Surgery
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Erin Duecy, Associate Professor, University of Rochester
Other Study IDs: 25003
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-05

CONDITIONS: Urogynecology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to establish normal postoperative changes in blood pressure in women undergoing scheduled gynecologic surgery requiring inpatient postoperative care. Also, to establish if there is a difference in normal postoperative blood pressure changes between elderly and non-elderly women undergoing scheduled gynecologic surgery requiring inpatient postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent scheduled gynecologic surgery requiring inpatient postoperative care between January 2007 - January 2008

Exclusion Criteria:

* Women who experienced myocardial infarction, cardiac arrest or failure, pulmonary embolism, infection requiring intravenous antibiotics, intra- or postoperative hemorrhage requiring blood transfusion, renal failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gynecologic patients
Sampling Method: Non-Probability Sample
Enrollment: 528 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Duecy, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a chart review study. 37 participants were not analyzed because the data in their chart was not available.
Groups:
- Women Who Underwent Gynecologic Surgery: All women who underwent inpatient Gynecologic surgery between Jan 2007 and 2008.
Period: Overall Study
Arm/Group | Women Who Underwent Gynecologic Surgery
Started | 491
Completed | 491
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This was a chart review study. 37 participants were not analyzed because the data in their chart was not available.
Groups:
- Women Who Underwent Gyneologic Surgery: All women who underwent inpatient Gynecologic surgery between Jan 2007 and 2008.
Arm/Group | Women Who Underwent Gyneologic Surgery
Number analyzed (Participants) | 491
Age, Continuous [Mean (Full Range); unit: years] | 50 [22 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 491
  Male | 0
Region of Enrollment [Number; unit: participants] — This was a chart review study. 37 participants were not analyzed because the data in their chart was not available.
  participants
    United States | 491
Postmenopausal [Number; unit: participants] | 169
Hypertension [Number; unit: participants] | 163
Diabetes [Number; unit: participants] | 26
Gastroesophageal Reflux Disease [Number; unit: participants] | 185
depression/anxiety [Number; unit: participants] | 159

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Underwent Gynecologic Surgery
Description: 491 women were included in analysis. Measure is categorized by the type of surgery.
Time Frame: January 2007 to January 2008
Population: 491 women were included in analysis.
Measure: Number; unit: percentage of participants
Groups:
- Women Who Underwent Scheduled Gynecologic Surgery: All women who underwent inpatient Gynecologic surgery between Jan 2007 and 2008. Measure is categorized by the type of surgery.
Arm/Group | Women Who Underwent Scheduled Gynecologic Surgery
Number analyzed (Participants) | 491
percentage of participants
  abdominal | 42
  laparoscopic | 32
  vaginal | 26

2. Secondary Outcome: Percentage of Women With Asymptomatic Hypotension
Description: % women with asymptomatic hypotension
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Groups:
- Women Who Underwent GYN Surgery: All women who underwent inpatient GYN surgery between Jan 2007 and 2008.
Arm/Group | Women Who Underwent GYN Surgery
Number analyzed (Participants) | 491
percentage of participants
  < 65 years of age | 22.8
  65 years or older | 17.7

3. Secondary Outcome: Percentage of Participants Undergoing Different Types of Anesthesia
Description: Patients were given either general, regional or local-modified anesthesia care (LO-MAC). Some of the patients ended up getting both general and regional anesthesia (sometimes anesthesia team decides to add regional for postop pain control).
Time Frame: January 2007 to January 2008
Measure: Number; unit: percentage of participants
Arm/Group | Women Who Underwent Gynecologic Surgery
Number analyzed (Participants) | 491
percentage of participants
  general | 92
  local | 4
  LO-MAC | 6

4. Secondary Outcome: Surgical Time
Description: Length of surgery
Time Frame: January 2007 to January 2008
Measure: Mean (Full Range); unit: minutes
Arm/Group | Women Who Underwent Gynecologic Surgery
Number analyzed (Participants) | 491
minutes | 146 [12 to 420]

ADVERSE EVENTS:
Description: This was a retrospective chart review. Adverse events were not collected.
Arm/Group | Women Who Underwent Gynecologic Surgery
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No